CLINICAL TRIAL: NCT02226978
Title: An Open-label One-sequence Cross-over Pharmacokinetic Interaction Study of Steady-state Tipranavir/Ritonavir 500/200 mg With Single-dose Valaciclovir (500 mg) in Healthy Volunteers
Brief Title: Pharmacokinetic Interaction Study of Steady-state Tipranavir/Ritonavir (TPV/r) With Single-dose Valaciclovir (VAL) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1182.104
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Valacyclovir

ARMS (1):
- TPV/r with valaciclovir (Experimental): VAL 2 days (on days 1 and 13), TPV/r 12 days (on days 2 to 13)
  Interventions: Drug: Tipranavir; Drug: Ritonavir; Drug: Valaciclovir

INTERVENTIONS:
Drug: Tipranavir
Drug: Ritonavir
Drug: Valaciclovir

SUMMARY:
Assessment of the interaction of tipranavir/ritonavir (TPV/RTV) and valaciclovir (VAL), a prodrug of aciclovir (ACV)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and non-pregnant, non-lactating female subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and willingness to comply with all study requirements
* Age >19 and <59 years (20 - 58 years inclusive)
* Weight ≥ 60 kg
* Body mass index (BMI) >18.5 and <29.9 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Atrioventricular (AV) block including 1°
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hematological, oncological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Relevant history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Known hypersensitivity to TPV, RTV, valaciclovir, aciclovir or antiretroviral drugs (marketed or experimental use as part of clinical research studies)
* Known elevated liver enzymes in past trials with any compound
* Intake of drugs with a long half-life (>24 hours) (<1 month prior to administration)
* Prescription or over the counter medications (including vitamins, minerals, herbal supplements and antacids), dietary supplements 14 days prior to study drug administration or expected during the trial)
* Participation in another trial with an investigational drug (<2 months prior to administration or expected during trial)
* Smoker with a consumption of >10 cigarettes or >3 cigars or >3 pipes/day and those who cannot keep tobacco intake constant
* Alcohol (>40 g/day for males and >20 g/day for females) and drug abuse
* Blood donation or loss >400 mL, < 3 month prior to administration
* Clinically relevant laboratory abnormalities
* Transaminases above reference values in the history
* Inability to comply with dietary regimen of study centre

For female subjects:

* Pregnancy or planning to become pregnant within 60 days of study completion
* Positive pregnancy test
* Have not been using a barrier method of contraception for at least 3 months prior to participation in the study if of childbearing potential and not surgically sterilized
* Are not willing or are unable to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during and up to 2 months after completion/termination of the trial if of childbearing potential and not surgically sterilized
* Chronic use of oral contraception or hormone replacement containing ethinyl estradiol
* Breast-feeding

Ages: 20 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of aciclovir in plasma over the time interval t0h to t12h (AUC0-12) | up to 12 hours after drug administration
Maximum measured concentration of aciclovir in plasma (Cmax) | up to 12 hours after drug administration

SECONDARY OUTCOMES:
AUC0-12 for Tipranavir (TPV) | up to 12 hours after drug administration
Cmax for TPV | up to 12 hours after drug administration
Drug concentration of TPV in plasma at 12 hours after administration (C12h) | up to 12 hours after drug administration
Apparent clearance of the analyte in the plasma after extravascular administration (CL/F) | up to 12 hours after drug administration
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | up to 12 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | up to 12 hours after drug administration
Number of subjects with adverse events | up to 14 days after last drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 14 days after last drug administration
AUC0-12 for Ritonavir (RTV) | up to 12 hours after drug administration
Cmax for RTV | up to 12 hours after drug administration
Drug concentration of RTV in plasma at 12 hours after administration (C12h) | up to 12 hours after drug administration